CLINICAL TRIAL: NCT00839709
Title: Peripheral Immunologic Response of Solid Organ Transplant Recipients to Depletion vs. Non-depletion Protocols
Brief Title: Peripheral Immunologic Response of Solid Organ Transplant Recipients to Depletion Versus Non-depletion Protocols
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Jorge Reyes, M.D., University of Washington
Other Study IDs: 34710-B
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Liver Disease; Liver Transplantation
Keywords: liver disease; liver transplantation; depletion immunosuppression; non-depletion immunosuppression
MeSH Terms: conditions — Liver Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- depletion immunosuppression
  Interventions: Procedure: blood sampling
- no depletion immunosuppression
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — peripheral blood draw

SUMMARY:
Rejection and infection are primary causes of morbidity and mortality in solid organ transplant recipients. Current clinical practice relies on immunosuppressive drug levels measured in plasma to reflect the peripheral immune response in solid organ transplant recipients. Direct measurement of the number and functions of the immune cells themselves using multi-parameter flow cytometry may enable individualized immunosuppression management for organ transplant recipients. Multi-parameter flow cytometry will be used to compare levels and functional capabilities of multiple lymphocyte subsets between cohorts of patients receiving depletion induction and those receiving a non-depletion regimen. The activation state, cytotoxic potential and the functional capabilities of these cells will be examined within patients over the first six months post transplant.

ELIGIBILITY:
Inclusion Criteria:

* liver transplant recipient

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge D Reyes, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States